CLINICAL TRIAL: NCT03253510
Title: Comparison Between Biting Force of Heat Cured Poly Methylmethacrylate and Metal Reinforced Polyamide for Mandibular Complete Denture
Brief Title: Measuring Biting Force of Poly-amide Complete Dentures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Hadi, Master degree candidate at removable prosthodontic department, Cairou, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Poly-amide complete dentures
Record Dates: First submitted 2017-08-10; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Complete Edentulism
MeSH Terms: interventions — Nylons; Polymethyl Methacrylate

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two more groups in parallel for the duration of the study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Poly-amide (Experimental): new thermoplastic material used as a denture base, that has excellent ethetics and flexibility
  Interventions: Other: Poly-amide
- poly-methyl methacrylate (Active Comparator): Polymethylmethacrylate is one of the most widely used denture base material, because of its good biocompatibility, reliability and dimensional stability
  Interventions: Other: Poly-methyl methacrylate

INTERVENTIONS:
Other: Poly-amide — New denture base material that exhibit high flexibility, physical strength, heat and chemical resistance and the exceedingly rare allergy response
  Other Names: Nylon
  Arms: Poly-amide
Other: Poly-methyl methacrylate — Gold standard denture base material
  Other Names: PMMA
  Arms: poly-methyl methacrylate

SUMMARY:
Randomized clinical trial to compare between biting force of mandibular complete denture constructed from two different materials; metal reinforced polyamide and conventional PMMA,The null hypothesis of the study that there will not be a difference between biting force of the complete denture constructed from metal reinforced polyamide and PMMA

DETAILED DESCRIPTION:
Polyamide resins used in dentistry exhibit high flexibility, physical strength, heat and chemical resistance and the exceedingly rare allergy response. Although flexural strength, modulus of elasticity and rigidity of nylon (polyamide) denture base materials are relatively low, they demonstrate great impact strength, toughness, and resistance to fracture. It was suggested that by adding glass fibers to polyamides, their stiffness and other mechanical properties could be increased. The flexural properties of nylon denture base materials has promoted their usage only in conditions like unyielding undercuts, pronounced tuberosities, tori and bulging alveolar ridges. In 2013 Wadachi etal compared rigidity of polyamide and PMMA when used as a denture base material and concluded that; the modulus of elasticity of polyamide was very low in comparison to PMMA and was lower than ISO standard, and so they recommended that polyamide to be used as a denture base material it should be reinforced with metal frame

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient with age range from fifty five to sixty five completely edentulous and in good medical condition
2. Patients have skeletal Angle's class I maxillo-mandibular relationship and sufficient inter arch distance.
3. Free from any systemic or neuromuscular disorder that might affect chewing efficiency of masticatory muscles.
4. Free from any tempro-mandibular disease.
5. Good oral hygiene

Exclusion Criteria:

1. Neuromuscular disorder and orofacial disease.
2. Tempromandibular joint and muscle pain
3. xerostomia or excessive salivation.
4. Limited mouth opening
5. Abnormal tongue behavior and/or size.
6. Intraoral soft and hard tissue pathosis

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Biting force | One month
  Bite force will be measured for both types of complete denture after one month of denture insertion . The recorded force during maximal clenching was obtained with I-load sensor placed between pairs of opposing teeth at one side and wood tongue depressor at the other side. The meter and depressor were located at the area of premolar/molar where there is more number of occlusal contacts with strong determinant of muscle action and subsequent great bite force.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadeer Hadi, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided